CLINICAL TRIAL: NCT04833777
Title: Does Addition of Longer-acting Local Anesthetic Improve the Post-operative Pain After Carpal Tunnel Release? A Randomized Controlled Study
Brief Title: Does a Different Local Anesthetic Improve Pain After Carpal Tunnel Release?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon City Hospital (Other)
Responsible Party: Principal Investigator, David Sauder, Principal Investigator, orthopedic surgeon, University of Saskatchewan
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Bio2640
Record Dates: First submitted 2021-03-26; First posted 2021-04-06 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: lidocaine; bupivacaine; carpal tunnel release
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Lidocaine, Prilocaine Drug Combination; Bupivacaine

STUDY DESIGN:
Intervention Model Description: The study model for the primary outcome will be single group (patients randomized to one of two anesthetic types). However, select patients who wish to have bilateral carpal tunnel release will be entered into a crossover model, such that they will be randomized for their first surgery and receive the other type of anesthetic for their second surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: The surgeon administering the local anesthetic will not be blinded, however the participant and the research nurse (measuring outcomes) will be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): Administration of subcutaneous lidocaine as local anesthetic prior to carpal tunnel release (lidocaine intervention)
  Interventions: Drug: Local Anesthetics Lidocaine
- Bupivacaine (Experimental): Administration of subcutaneous bupivacaine + lidocaine as local anesthetic prior to carpal tunnel release (bupivacaine intervention)
  Interventions: Drug: Local Anesthetics Bupivacaine

INTERVENTIONS:
Drug: Local Anesthetics Lidocaine — 10 mL 1% lidocaine with 1:100,000 epinephrine and 1 mL 8.4% sodium bicarbonate
  Arms: Lidocaine
Drug: Local Anesthetics Bupivacaine — 5 mL 1% lidocaine with 1:100,000 epinephrine + 5 mL 0.5% bupivacaine with 1:100,000 epinephrine and 1 mL 8.4% sodium bicarbonate
  Arms: Bupivacaine

SUMMARY:
This study is being conducted to determine whether addition of a longer-acting local anesthetic to our current anesthetic protocol improves the post-operative pain after carpal tunnel release. Participants undergoing carpal tunnel release (CTR) will be randomly assigned to one of two groups: the standard anesthetic or the longer-acting anesthetic. Participants will not be aware of their assignment. Carpal tunnel release will be performed in the standard fashion at our hospital. Participants will record their post-operative pain on a visual scale at 2, 4, 6, 8, and 10 hours after surgery. They will also record the location of their post-operative numbness at the same time intervals. The day after surgery, a research nurse will call each participant to inquire about their post-operative pain scores and numbness. Participants will also be asked about their consumption of oral painkillers (e.g. Tylenol, ibuprofen) during the first 24 hours. Participants will be re-assessed 3 months after surgery to evaluate improvement in carpal tunnel symptoms.

Participants who wish to have carpal tunnel release on both wrists will be randomized to receive one type of anesthetic for the first side and will receive the other anesthetic for the second side. They will not be made aware of which medication is used for each side. This will allow us to directly compare the difference in pain experience between the two anesthetics.

We hypothesize that use of a longer-acting local anesthetic will lead to decreased post-operative pain, especially in the first 4-8 hours after surgery.

DETAILED DESCRIPTION:
A research nurse will meet with each patient presenting for outpatient CTR surgery at the Saskatoon City Hospital procedure room. He or she will obtain informed consent for interested participants. The patient will be assigned a subject number and be randomized to standard vs. bupivacaine treatment based on a computer algorithm. Participants will complete the Boston Carpal Tunnel Questionnaire as a baseline for comparison as well as a brief questionnaire on demographics. For those patients that are having both sides released during the study period, the first side will be randomized based on the study protocol and the second side will be anesthetized with the other treatment. They will be blinded to both procedures such that we can directly compare their operative experience.

The surgeon will draw up and mix the pre-determined local anesthetic (LA) for each patient based on the randomization protocol. The research nurse (who will be performing all assessments) and the patient will remain blinded to the type of anesthetic.

The two types of anesthetic will be:

1. 10 mL 1% lidocaine with 1:100,000 epinephrine and 1 mL 8.4% sodium bicarbonate (standard treatment)
2. 5 mL 1% lidocaine with 1:100,000 epinephrine + 5 mL 0.5% bupivacaine with 1:100,000 epinephrine and 1 mL 8.4% sodium bicarbonate (bupivacaine treatment)

The participants will be anesthetized in the standard fashion, with all 11 mL of LA infiltrated subcutaneously into the area of the incision. After a delay of 20-40 minutes, the CTR will be carried out using the standard mini-open approach. Patients will be provided with the standard post-operative instructions regarding activity and wound care.

After the procedure, participants will complete a short questionnaire (VAS) about any pain experienced during the administration of the local anesthetic and during the procedure. Patients will be sent home with instructions to complete a pain and numbness assessment at 2, 4, 6, 8, and 10 hours after surgery. They will be provided with a form containing the VAS and the times at which they are to self-administer this pain scoring system. Additionally, they will be provided with 20 Tylenol tablets (325mg each) and 20 ibuprofen tablets (200mg each), with instructions to take 1-2 tablets of one or both analgesics every 6 hours as needed during the first 24 hours. They will be asked to document the times at which they took the medications, as well as the dosages taken. They will be asked to refrain from using other types of pain medications, if possible. They will also be asked to document use of any other analgesics including Cannabis. Any questions will be answered by the research nurse before leaving clinic.

The day after surgery, at the 24 hour mark, the research nurse will call each patient and inquire about their pain scores and numbness at 2, 4, 6, 8, and 10 hours, as well as the present time (24 hours). He or she will also ask about the number of Tylenol and/or ibuprofen pills taken during the first 24 hours, as well as the timing of consumption. This information recorded on a password-protected datasheet which contains only the subject number (no identifiers).

The patient will return for their standard follow-ups. At 3 months, the research nurse will repeat the Boston Carpal Tunnel Questionnaire to assess outcome. At this time, if the patient wishes, they may be unblinded.

For patients wishing for bilateral CTR, the first will be performed according to the randomization protocol as described above. The contralateral CTR will be performed 2-8 weeks later (as standard in our practice), with the alternate anesthetic (e.g. first CTR with standard treatment, second CTR with bupivacaine treatment). The same post-operative assessment will be performed for the second CTR. Patients will remain blinded to their type of anesthetic in each wrist until 3 months after the second surgery is performed. At that time, they will be asked by the research nurse whether the first or second surgery provided a better pain experience. Only after this will they be unblinded, if desired.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years undergoing carpal tunnel release

Exclusion Criteria:

* Patients aged <18 years
* Patients undergoing repeat carpal tunnel release
* Patients undergoing simultaneous procedures for other hand/wrist pathology at the time of carpal tunnel release (i.e. trigger finger release, Dupuytren's, etc.)
* Patients with a history of Rheumatoid Arthritis or a history or previous trauma or surgery to the local area (i.e. distal radius fracture)
* Patients who lack the capacity to provide informed consent or understand the nature of the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sauder, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Saskatoon City Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Wrist
Period: Overall Study
Arm/Group | Lidocaine | Bupivacaine
Started (While units are the number of wrists that had carpal tunnel release, each participant was only enrolled once. E.g. a patient who was randomized during surgery of their right wrist, would not be enrolled again if they returned for surgery on their left wrist.) | 68; 68 Wrist | 72; 72 Wrist
Data Analysis | 67; 67 Wrist | 72; 72 Wrist
Completed | 67; 67 Wrist | 72; 72 Wrist
Not Completed | 1; 1 Wrist | 0; 0 Wrist
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Bupivacaine | Total
Number analyzed (Participants) | 67 | 72 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.9) | 63 (16.6) | 60 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 35 | 62
  Male | 40 | 37 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 67 | 72 | 139

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: Severity of pain as measured by the Visual Analogue Scale. This tool asks patients to rate their post-operative pain level from 0 to 10. 0 represents no pain, while 10 represents the worst possible pain.
Time Frame: 2 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (Wrists) | 67 | 72
score on a scale | 1.16 (1.83) | 0.92 (1.61)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 4 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (Wrists) | 67 | 72
score on a scale | 2.16 (2.23) | 1.54 (1.98)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 6 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
score on a scale | 3.19 (2.29) | 2.29 (2.35)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 8 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
score on a scale | 3.87 (2.24) | 2.92 (2.30)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 10 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
score on a scale | 3.81 (2.32) | 3.38 (2.42)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 24 hours post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
score on a scale | 3.22 (2.22) | 3.38 (2.35)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Post-operative Analgesia Requirements
Description: Number of Tylenol and Ibuprofen tablets taken post-operatively within the first 24 hours. This was not measured on a scale. Patients were asked to count the total number of Tylenol (500mg) and Ibuprofen (200mg) tablets they consumed within the first 24 hours after surgery.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: number of tablets
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
number of tablets | 7.45 (4.70) | 7.31 (4.57)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Post-operative Analgesia Requirements
Description: Number of Tylenol and Ibuprofen tablets taken post-operatively within the first 24 hours. This was not measured on a scale. Patients were asked to count the total number of Tylenol (500mg) and Ibuprofen (200mg) tablets they consumed within the first 72 hours after surgery.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: number of tablets
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
number of tablets | 14.5 (11.8) | 13 (8.9)
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Post-operative Numbness
Description: Presence of post-operative numbness in any finger (thumb, index, middle, ring, or little finger). Patients answer "yes" or "no" to numbness.
Time Frame: 2 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 55 | 58
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

10. Secondary Outcome: Post-operative Numbness
Description: as for outcome 9
Time Frame: 4 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 55 | 64
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

11. Secondary Outcome: Post-operative Numbness
Description: as for outcome 9
Time Frame: 6 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 43 | 63
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

12. Secondary Outcome: Post-operative Numbness
Description: as for outcome 9
Time Frame: 8 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 31 | 59
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

13. Secondary Outcome: Post-operative Numbness
Description: as for outcome 9
Time Frame: 10 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 21 | 51
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

14. Secondary Outcome: Post-operative Numbness
Description: as for outcome 9
Time Frame: 24 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 17 | 33
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

15. Secondary Outcome: Symptom Change at 3 Months
Description: Carpal tunnel symptoms at 3 months post-op, measured by the Boston Carpal Tunnel Questionnaire. The BCTQ is a self- administered questionnaire consisting of two domains: a symptom severity scale (SSS) and a functional status scale (FSS). Each item on the questionnaire is scored on a 5-point rating scale, with higher scores indicating greater disability. The symptom severity scale ranges from 11 to 55, and the functional status scale ranges from 8 to 40, with higher scores indicating greater disability.
Time Frame: pre-operative/baseline (immediately before surgery), 3 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wrists
Groups:
- Lidocaine-baseline BCTQ SSS; Lidocaine-baseline BCTQ FSS; Lidocaine-3 Months Post-op BCTQ SSS; Lidocaine-3 Months Post-op BCTQ FSS: Administration of subcutaneous lidocaine as local anesthetic prior to carpal tunnel release (lidocaine intervention)
  Local Anesthetics Lidocaine: 10 mL 1% lidocaine with 1:100,000 epinephrine and 1 mL 8.4% sodium bicarbonate
- Bupivacaine-baseline BCTQ SSS; Bupivacaine-baseline BCTQ FSS; Bupivacaine-3 Months Post-op BCTQ SSS; Bupivacaine-3 Months Post-op BCTQ FSS: Administration of subcutaneous bupivacaine + lidocaine as local anesthetic prior to carpal tunnel release (bupivacaine intervention)
  Local Anesthetics Bupivacaine: 5 mL 1% lidocaine with 1:100,000 epinephrine + 5 mL 0.5% bupivacaine with 1:100,000 epinephrine and 1 mL 8.4% sodium bicarbonate
Arm/Group | Lidocaine-baseline BCTQ SSS | Lidocaine-baseline BCTQ FSS | Bupivacaine-baseline BCTQ SSS | Bupivacaine-baseline BCTQ FSS | Lidocaine-3 Months Post-op BCTQ SSS | Lidocaine-3 Months Post-op BCTQ FSS | Bupivacaine-3 Months Post-op BCTQ SSS | Bupivacaine-3 Months Post-op BCTQ FSS
Number analyzed (Participants) | 67 | 67 | 72 | 72 | 67 | 67 | 72 | 72
Number analyzed (wrists) | 67 | 67 | 72 | 72 | 67 | 67 | 72 | 72
score on a scale | 33.1 (7.1) | 19.6 (6.4) | 34.5 (7.1) | 20.7 (6.4) | 15.3 (5.9) | 10.5 (3.8) | 15 (4.7) | 10.8 (3.7)

16. Secondary Outcome: Post-operative Numbness
Description: as for outcome 9
Time Frame: 48 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 13 | 26
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

17. Secondary Outcome: Post-operative Numbness
Description: as for outcome 9
Time Frame: 72 hours post-op
Measure: Count of Units; unit: wrists
Units Other Than Participants: wrists
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 67 | 72
Number analyzed (wrists) | 67 | 72
wrists | 10 | 24
Statistical Analysis 1: Comparison: Lidocaine vs Bupivacaine; Test type: Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Lidocaine | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/72
Other Adverse Events (participants affected / at risk) | 0/67 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04833777/Prot_SAP_000.pdf